CLINICAL TRIAL: NCT06233539
Title: A Study on Diagnosis and Treatment Strategies for Atlantoaxial Dislocation
Status: Recruiting | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2022822
Record Dates: First submitted 2024-01-22; First posted 2024-01-31 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-01

CONDITIONS: Atlantoaxial Dislocation; Treatment; Diagnostic
MeSH Terms: conditions — Disease | interventions — Methods

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective section
  Interventions: Other: Observational research without intervention
- Prospective section
  Interventions: Other: Observational research without intervention

INTERVENTIONS:
Other: Observational research without intervention — Observational research without intervention

SUMMARY:
The most effective treatment for atlantoaxial dislocation is surgical treatment, with the principle of achieving reduction, reconstruction, and fusion of the atlantoaxial joint. The surgical strategies mainly include simple anterior approach, simple posterior approach, and combined anterior posterior approach. The investigators have summarized 904 cases of atlantoaxial instability or dislocation from 1998 to 2010 and preliminarily published the diagnosis and treatment strategy tree of the Third Hospital of Beijing Medical University. This strategy is divided into four types based on the severity of atlantoaxial dislocation: unstable, reversible, difficult to recover, and skeletal, and enters different surgical treatment processes. With the increase in the number of cases, accumulation of experience, and technological improvements in the past decade, spinal surgery colleagues have updated their classification diagnosis, diagnosis and treatment processes, and surgical techniques for atlantoaxial instability or dislocation.

However, the selection of treatment strategies for atlantoaxial dislocation is mostly based on the surgeon's own experience, and there is a lack of standardized, large-scale, and high-level evidence-based medical research on the safety and effectiveness of current empirical strategies. Based on this, this study intends to adopt a multicenter, retrospective, and prospective study to construct a high-quality clinical cohort of atlantoaxial dislocation, update the classification and diagnosis and treatment strategies of atlantoaxial dislocation. And conduct long-term follow-up on patients to evaluate their safety and effectiveness, guide the surgical treatment of atlantoaxial dislocation, and thus form a recognized diagnostic and treatment standard for atlantoaxial dislocation.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with atlantoaxial dislocation and treated with surgery

Exclusion Criteria:

* Disagree to participate in this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with atlantoaxial dislocation and treated with surgery
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of special attention adverse events in patients within 12 months after surgery | 12 month follow up
  The proportion of adverse events occurring in patients during the study period to the total number of study patients.
  Recording and reporting of adverse events, including: • deterioration of neurological function
  * Incision infection
  * Vascular injury
  Airway obstruction
  Poor reset
  • Unplanned readmission and unplanned reoperation • Internal fixation failure
  Fusion failure
  Surgical related lower cervical spine deformities

CONTACTS AND LOCATIONS:
Locations (1):
- Shenglin Wang, Beijing, Beijing Municipality, China